CLINICAL TRIAL: NCT04098770
Title: Safety and Efficiency of Allogeneic Adoptive Immune Therapy for Advanced AIDS Patients
Brief Title: Allogeneic Adoptive Immune Therapy for Advanced AIDS Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing 302 Hospital (Other)
Collaborators: The 6th people's Hospital of Xinjiang province (Unknown); The 4th people's hospital of Nanning City (Unknown); The 3th people's hospital of Shenzhen City (Unknown); Shanghai Public Health Clinical Center (Other Government); Yunnan Provincial Hospital of Infectious Diseases (Unknown)
Responsible Party: Principal Investigator, Fu-Sheng Wang, Head of Treatment and Research Center for Infectious Diseases, Principle Investigator, Clinical Professor, Beijing 302 Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 302-2019-05
Record Dates: First submitted 2019-08-29; First posted 2019-09-23 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-06

CONDITIONS: AIDS Patients
Keywords: AIDS patients; Safety; Efficiency; Immune Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional treatment plus Allogeneic Adoptive Immune Therapy (Experimental): Participants will receive conventional treatment (anti-opportunistic infections, cART and other treatments) plus a dose (2-3 times) of Allogeneic Adoptive Immune Therapy
  Interventions: Biological: Allogeneic Adoptive Immune Therapy
- Conventional treatment (No Intervention): Without Allogeneic Adoptive Immune Therapy but conventional treatment (anti-opportunistic infections , cART and other treatments) should be received

INTERVENTIONS:
Biological: Allogeneic Adoptive Immune Therapy — A dose (2-3 times) of AAIT was added on conventional treatment for advanced AIDS patients
  Arms: Conventional treatment plus Allogeneic Adoptive Immune Therapy

SUMMARY:
Combined antiretroviral therapy (ART) efficiently suppresses viral replication and markedly decreases mortality among patients with HIV-1 infection/AIDS. While the advanced AIDS patients with CD4+T cell count less than 200 cells/µL often develop seriously opportunistic infections (OIs), severe wasting syndrome, and other fatal complications, which are the major causes of death in these patients. There has been no effective immune therapy for advanced AIDS patients who had a high mortality rate even in the era of cART. This clinical trail is to inspect the efficiency of allogeneic adoptive immune therapy for advanced AIDS patients.

DETAILED DESCRIPTION:
Combined antiretroviral therapy (ART) efficiently suppress viral replication and dramatically decrease mortality of the disease in HIV-1/AIDS patients.1 While in cART naive patients with chronic human immunodeficiency virus-1 (HIV-1) infection often characterized by HIV-1 replication, immune activation and deficiency, which lead to profound and systematic inflammation and pathoglogical change, especially in the AIDS patients with CD4 T count less than 50/uL, who often develop deadly complications, which accounts for the major cause of death group in spite of cART era. Up-to-date, there are no effective immune interventions to restore host holistic immunity for advanced AIDS patients.

In pre-cARTera, HLA-matched lymphocytes or stem cell transplantation had been exploratively used in AIDS patients. However, this kind of therapy failed for immunological reconstitution due to the lack of antiviral therapy to suppress HIV-1 replication at that time. With the advent of cART, allogeneic HLA-matched or mismatched lymphocytes or stem cell transplantations were mainly used for AIDS patients with hematopoietic malignancies, the Berlin and London patients were the cured pateints. However, allogeneic transplantation can not be used outside the setting of hematopoietic malignancies. In addition, the high frequency of GVHD (Graft-versus-host disease) owning to a transient or long-lasting engraftment is inevitable.

Until now, there has been no report of effective immune therapy for late-stage AIDS patients with acquired immunodeficiency and severe opportunistic infections (OIs). The urgent challenge is how to efficiently restore the host holistic immunity in AIDS patients at late stage.

The investigators have recently developed a mismatched allogeneic adoptive immune therapy (AAIT) protocol in combination with cART, and found that the treatment was safety and tolerability in a phase I study. The purpose of this study is to further investigate the efficacy of allogeneic adoptive immune therapy (AAIT) for advanced AIDS patients. 120 patients received i.v. transfusion one round (2-3 times) of 1.0-3.0*10E8 cells/kg of MNSs as the treated group, all of these patients received the conventional cART treatment. In addition, the equal 120 patients received cART were used as control. The side effects, CD4 T cell numbers, HIV viral load, clinical symptoms improvement, control of opportunistic infections, AIDS-related events and non-AIDS related events will be evaluated during the 96-week follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged at 18 years (including) -65 years old
2. Advanced AIDS patients with AIDS-related events
3. Advanced patients with CD4 count less than or equal to 200 cells/uL, including end-stage patients with CD4 count less than or equal to 50 cells/uL before entry and at screening
4. Sign informed consent, do not participate in other clinical trails during the period

Exclusion Criteria:

1. Pregnancy, lactation and those who are not pregnant but do not take effective contraceptives measures
2. Combined with other serious organic diseases while didn't related with AIDS
3. HIV-2 infection
4. Allergic to blood products
5. Under long term immunosuppressive therapy
6. Combined with malignant tumors
7. Drug addicts within half-one year before the test
8. Poor compliance to antiviral therapy; take part in other clinical trials at present

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2019-10-11 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
The change of CD4+ T cell count between AAIT treatment group and conventional group | At Baseline , week 4,12, 24, 48 and 96
  Marker for host immunity
The change of survival between AAIT treatment group and conventional group | At week 24, 48 and 96
  Marker for efficacy of treatment

OTHER OUTCOMES:
Side effects in the AAIT treatment group | At Baseline, week 1, 2 , 4 and 24
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
The occurence of clinical events including AIDS-related events and non-AIDS related events in the two groups | At baseline, week 24, 48, 84 and 96
  Marker for efficacy of treatment
The change of plasma RNA copies/mL between AAIT treatment group and conventional group | At Baseline, week 1, 4, 12, 24, 48, 84 and 96
  Marker for HIV viral load
The change of plasma HIV DNA between AAIT treatment group and conventional group | At Baseline and week 1, 12, 24 and 48
  Changes of HIV DNA in PBMC

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Sheng Wang, MD, Study Director — Beijing 302 Hospital
Locations (1):
- Beijing 302 Hospital of China, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kuritzkes DR. Hematopoietic stem cell transplantation for HIV cure. J Clin Invest. 2016 Feb;126(2):432-7. doi: 10.1172/JCI80563. Epub 2016 Jan 5. PMID 26731468
- [Background] Hutter G, Nowak D, Mossner M, Ganepola S, Mussig A, Allers K, Schneider T, Hofmann J, Kucherer C, Blau O, Blau IW, Hofmann WK, Thiel E. Long-term control of HIV by CCR5 Delta32/Delta32 stem-cell transplantation. N Engl J Med. 2009 Feb 12;360(7):692-8. doi: 10.1056/NEJMoa0802905. PMID 19213682
- [Background] Krishnan A. Stem cell transplantation in HIV-infected patients. Curr Opin HIV AIDS. 2009 Jan;4(1):11-5. doi: 10.1097/COH.0b013e32831a6fc9. PMID 19339935
- [Background] Davis KC, Hayward A, Ozturk G, Kohler PF. Lymphocyte transfusion in case of acquired immunodeficiency syndrome. Lancet. 1983 Mar 12;1(8324):599-600. doi: 10.1016/s0140-6736(83)92855-6. No abstract available. PMID 6131294
- [Background] Lane HC, Masur H, Longo DL, Klein HG, Rook AH, Quinnan GV Jr, Steis RG, Macher A, Whalen G, Edgar LC, et al. Partial immune reconstitution in a patient with the acquired immunodeficiency syndrome. N Engl J Med. 1984 Oct 25;311(17):1099-103. doi: 10.1056/NEJM198410253111706. No abstract available. PMID 6384784
- [Background] Lane HC, Zunich KM, Wilson W, Cefali F, Easter M, Kovacs JA, Masur H, Leitman SF, Klein HG, Steis RG, et al. Syngeneic bone marrow transplantation and adoptive transfer of peripheral blood lymphocytes combined with zidovudine in human immunodeficiency virus (HIV) infection. Ann Intern Med. 1990 Oct 1;113(7):512-9. doi: 10.7326/0003-4819-113-7-512. PMID 1975487
- [Derived] Yang T, Xie Z, Xu Z, Tu B, Lu H, Huang H, Huang L, Zhang C, Gao L, Jin L, Ma P, Zou J, Liu L, Zhen C, Zhou C, Meng S, Li YY, Song JW, Yang S, Ai HS, Jiao Y, Shi M, Xu R, Wang FS. HLA-mismatched allogeneic adoptive immune therapy in patients with severely immunosuppressed AIDS: a multicenter, open-label, controlled, phase 2a study. Emerg Microbes Infect. 2024 Dec;13(1):2364744. doi: 10.1080/22221751.2024.2364744. Epub 2024 Jun 27. PMID 38935839